CLINICAL TRIAL: NCT01101542
Title: Safety of GlaxoSmithKline (GSK) Biologicals' Human Papillomavirus (HPV)-16/18 Vaccine, Cervarix® When Administered to Healthy Females According to the Prescribing Information in Korea
Brief Title: Evaluation of Safety of a Vaccine Against Cervical Cancer in Healthy Korean Females
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112485
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2015-10

CONDITIONS: Infections, Papillomavirus
Keywords: Post-marketing surveillance; Human papillomavirus; Korea; Safety; Prescribing Information
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cervarix Group: Subjects received 3 doses of the Cervarix vaccine. The vaccine was administered intramuscularly into the deltoid muscle of the non-dominant arm according to a 0,1, 6 month vaccination schedule. According to the prescribing information, if flexibility in the vaccination schedule is necessary, the second dose can be administered between 1 month and 2.5 months after the first dose.
  Interventions: Biological: Cervarix.; Other: Data collection

INTERVENTIONS:
Biological: Cervarix. — Subjects will receive three doses of the Cervarix vaccine administered intramuscularly according to a 0, 1, 6 month vaccination schedule in routine clinical practice settings.
Other: Data collection — All adverse events will be recorded by all subjects or the subject's parents/guardians using diary cards.

SUMMARY:
This Post Marketing Surveillance (PMS) will collect safety data on the use of GSK Biologicals' human papillomavirus (HPV) vaccine in the local target population of females as per the regulations of the Korean Food and Drugs Administration (KFDA).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged between and including, 10 to 25 years at the time of the first vaccination.
* Subjects who the investigator believes that they or their parents/guardians can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for vaccination visits etc) should be enrolled in the PMS.
* Written informed consent obtained from the subject or the subjects' parent/ guardian.
* Subjects of childbearing potential must not be pregnant. Absence of pregnancy should be verified (e.g. urine pregnancy test) as per the investigator's clinical judgement.
* Subjects with no contraindication according to the local approved prescribing information.
* No previous administration of an HPV vaccine other than Cervarix®.
* No previous administration of more than two doses of Cervarix®.
* No planned administration of an HPV vaccine other than Cervarix® during the PMS

Ages: 10 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy female subjects aged between and including 10 to 25 years who receive Cervarix® according to the current practice of Korean doctors.
Sampling Method: Non-Probability Sample
Enrollment: 3091 (Actual)
Dates: Start 2010-07-01; Primary Completion 2014-02-20 (Actual); Study Completion 2014-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- South Korea (2):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Seoul

REFERENCES:
- [Derived] Kim CJ, Song R, Chen J, Tavares Da Silva F, Gopala KB, Kim JH, Bi D, Park JS. Six-year multi-centre, observational, post-marketing surveillance of the safety of the HPV-16/18 AS04-adjuvanted vaccine in women aged 10-25 years in Korea. Pharmacoepidemiol Drug Saf. 2017 Jul;26(7):837-842. doi: 10.1002/pds.4175. Epub 2017 Mar 7. PMID 28266092

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As per study protocol, subjects who had received 1 or 2 doses of Cervarix vaccine prior to the start of the Post-Marketing Surveillance Study (PMS) could also be enrolled. A total of 3091 participants were enrolled in the study, 105 were available for Year 3 Surveillance and 569 were available for Year 4 Surveillance.
Groups:
- Cervarix Group: Subjects who received 3 doses of the Cervarix vaccine. The vaccine was administered intramuscularly into the deltoid muscle of the non-dominant arm according to a 0,1, 6 month vaccination schedule. According to the prescribing information, if flexibility in the vaccination schedule was necessary, the second dose could be administered between 1 month and 2.5 months after the first dose.
Period: Year 3 Surveillance Period
Arm/Group | Cervarix Group
Started | 105
Completed | 94
Not Completed | 11
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 4
Period: Year 4 Surveillance Period
Arm/Group | Cervarix Group
Started | 569
Completed | 282
Not Completed | 287
Not completed — Other | 287
Period: Year 5 Surveillance Period
Arm/Group | Cervarix Group
Started | 809
Completed | 668
Not Completed | 141
Not completed — Lost to Follow-up | 140
Not completed — Pregnancy | 1
Period: Year 6 Surveillance Period
Arm/Group | Cervarix Group
Started | 3091
Completed | 2100
Not Completed | 991
Not completed — Lost to Follow-up | 986
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- Cervarix Group: Subjects received 3 doses of the Cervarix vaccine. The vaccine was administered intramuscularly into the deltoid muscle of the non-dominant arm according to a 0,1, 6 month vaccination schedule. According to the prescribing information, if flexibility in the vaccination schedule was necessary, the second dose could be administered between 1 month and 2.5 months after the first dose.
Arm/Group | Cervarix Group
Number analyzed (Participants) | 3091
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 3 of surveillance. Population: A total of 105 participants were included in the Year 3 surveillance.
  Years
    number analyzed (Participants) | 105
    (all) | 20.4 (3.72)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 4 of surveillance. Population: A total of 569 participants were included in the Year 4 surveillance.
  Years
    number analyzed (Participants) | 569
    (all) | 20.8 (3.87)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 5 of surveillance. Population: A total of 809 participants were included in the Year 5 surveillance.
  Years
    number analyzed (Participants) | 809
    (all) | 20.9 (3.06)
Age, Continuous [Mean (Standard Deviation); unit: Years] — The baseline measure data here corresponds to Year 6 of surveillance.
  Years | 20.5 (3.82)
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 3 of surveillance. Population: A total of 105 participants were included in the Year 3 surveillance.
  Participants
    number analyzed (Participants) | 105
    Female | 105
    Male | 0
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 4 of surveillance. Population: A total of 569 participants were included in the Year 4 surveillance.
  Participants
    number analyzed (Participants) | 569
    Female | 569
    Male | 0
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 5 of surveillance. Population: A total of 809 participants were included in the Year 5 surveillance.
  Participants
    number analyzed (Participants) | 809
    Female | 809
    Male | 0
Sex: Female, Male [Count of Participants; unit: Participants] — The baseline measure data here corresponds to Year 6 of surveillance.
  Participants
    Female | 3091
    Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 30-day period (Day 0 to Day 29) following any vaccination (During the 3rd year of surveillance).
Population: The analysis was performed on the Total Vaccinated cohort that included all vaccinated subjects with at least one dose of Cervarix vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 105
Subjects | 30

2. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
  Note: Results for the 5th and 6th year of surveillance will be added when they become available.
Time Frame: During the 30-day period (Day 0 to Day 29) following any vaccination (During the 4th year of surveillance).
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 569
Subjects | 88

3. Primary Outcome: Number of Subjects Reporting Serious Adverse Event (SAEs) and SAE(s) Causally Related to Vaccination.
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: During the entire Post Marketing Surveillance period up to one month after the third vaccine dose (During the 3rd year of surveillance).
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 105
Subjects
  Any SAEs | 0
  Related SAEs | 0

4. Primary Outcome: Number of Subjects Reporting Serious Adverse Event (SAEs) and SAE(s) Causally Related to Vaccination.
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
  Note: Results for the 5th and 6th year of surveillance will be added when they become available.
Time Frame: During the entire Post Marketing Surveillance period up to one month after the third vaccine dose (During the 4th year of surveillance).
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 569
Subjects | 2

5. Primary Outcome: Number of Subjects With Medically Significant Conditions.
Description: *Note: For Surveillance Year 3 the analysis was not performed for this outcome since it was not a requirement of the Korean regulatory authority.
Time Frame: During the entire Post Marketing Surveillance period up to one month after the third vaccine dose (During the 3rd, 4th, 5th and 6th year of surveillance)
Population: *Note: the analysis was not performed for this outcome since it was not a requirement of the Korean regulatory authority.
Arm/Group | Cervarix Group
Number analyzed (Participants) | 0

6. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: as for outcome 1
Time Frame: During the 30-day period (Day 0 to Day 29) following any vaccination (During the 5th year of surveillance).
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 809
Subjects | 214

7. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: as for outcome 1
Time Frame: During the 30-day period (Day 0 to Day 29) following any vaccination (During the 6th year of surveillance).
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 3091
Subjects | 620

8. Primary Outcome: Number of Subjects Reporting Serious Adverse Event (SAEs) and SAE(s) Causally Related to Vaccination.
Description: as for outcome 3
Time Frame: During the entire Post Marketing Surveillance period up to one month after the third vaccine dose (During the 5th year of surveillance).
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 809
Subjects
  Any SAEs | 2
  Related SAEs | 0

9. Primary Outcome: Number of Subjects Reporting Serious Adverse Event (SAEs) and SAE(s) Causally Related to Vaccination.
Description: as for outcome 3
Time Frame: During the entire Post Marketing Surveillance period up to one month after the third vaccine dose (During the 6th year of surveillance).
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 3091
Subjects
  Any SAEs | 3
  Related SAEs | 0

10. Primary Outcome: Number of Subjects With Medically Significant Conditions.
Description: MSC include AEs prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: During the entire Post Marketing Surveillance period up to one month after the third vaccine dose (During the 4th, 5th and 6th year of surveillance)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 3091
Subjects
  Subjects with any MSCs, Year 4 (N=569) | 27
  Subjects with any MSCs, Year 5 (N=809) | 44
  Subjects with any MSCs, Year 6 (N=3091) | 135

ADVERSE EVENTS:
Time Frame: Unsolicited AEs: During the 30-day period (Days 0-29) following any vaccination; SAEs: Throughout the PMS study period (up to one month after the third vaccine dose)
Description: Only adverse events with a frequency of over 5% were listed.
Groups:
- Cervarix Group: Subjects enrolled for surveillance Year 6, who received 3 doses of the Cervarix vaccine. The vaccine was administered intramuscularly into the deltoid muscle of the non-dominant arm according to a 0,1, 6 month vaccination schedule. According to the prescribing information, if flexibility in the vaccination schedule was necessary, the second dose could be administered between 1 month and 2.5 months after the first dose.
Arm/Group | Cervarix Group
Serious Adverse Events (participants affected / at risk) | 3/3091
Other Adverse Events (participants affected / at risk) | 322/3091
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=3091)
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=3091)
Injection site pain (General disorders) | 322

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.